CLINICAL TRIAL: NCT02509845
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Microbiology of C16G2 Administered in Multiple Oral Gel Doses to Adolescent and Adult Dental Subjects
Brief Title: Study to Evaluate the Safety and Microbiology of C16G2 in Adolescent and Adult Dental Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Armata Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C3J15-202-00
Record Dates: First submitted 2015-07-01; First posted 2015-07-28 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Antimicrobial Peptides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adolescent Safety Only Cohort (Experimental): Prior to commencing enrollment of subjects 12-17 years of age in Study Arms 1 & 2, a safety only cohort of 4 to 8 adolescent subjects will receive 4 administrations of C16G2 on Day 0.
  Interventions: Drug: C16G2; Other: Placebo
- Study Arm 1 (Experimental): Subjects will receive 2 mL of study drug or placebo over two 7 day C16G2 administration periods, which will be separated by approximately 4 months. Subjects enrolled in Study Arm 1 will receive 4 study drug or placebo administrations on the first day of dosing followed by morning (AM) and evening (PM) dosing for 6 consecutive days. Study drug will be administered via manual toothbrush and custom dental trays.
  Interventions: Drug: C16G2; Other: Placebo
- Study Arm 2 (Experimental): Subjects will receive 4 mL of study drug or placebo over two 7 day C16G2 administration periods, which will be separated by approximately 4 months. Subjects enrolled in Study Arm 2 will receive 4 study drug or placebo administrations on the first day of dosing followed by morning (AM) and evening (PM) dosing for 6 consecutive days. Study drug will be administered via manual toothbrush and custom dental trays.
  Interventions: Drug: C16G2; Other: Placebo

INTERVENTIONS:
Drug: C16G2 — Antimicrobial peptide
  Other Names: Antimicrobial peptide
Other: Placebo — Placebo

SUMMARY:
The purpose of the clinical study is to evaluate the safety and bacterial impact of study drug (C16G2) administered in multiple oral gel doses to adolescent and adult dental subjects.

DETAILED DESCRIPTION:
The purpose of the clinical study is to evaluate the safety and microbiology of C16G2 administered in multiple oral gel doses to adolescent and adult dental subjects. Subjects will be assigned to three study cohorts and receive 2 different volumes of C16G2 Gel or Placebo. Prior to commencing enrollment of subjects 12-17 years of age, a safety only cohort of 4-8 adolescent subjects will receive 4 study drug administrations on Day 0. A safety data review will be performed by the Medical Monitor on Days 1 and 5. If no safety concerns are identified, enrollment of adolescent subjects receiving 7 days of study drug administration will be initiated in Study Arms 1 & 2. Enrollment of adult subjects in Study Arms 1 & 2 may start before the Adolescent Safety Only Cohort is initiated. Before dosing of study drug, eligible subjects will undergo professional dental prophylaxis on Day 0. Microbiology will be assessed by measuring S. mutans and total bacteria counts.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent Safety Only Cohort: Males and females, 12-17 years of age, inclusive, at the time the Assent and Informed Consent Form is signed. Study Arms 1 & 2: Males and females, 12-75 years of age, inclusive, at the time the Assent and/or Informed Consent Form is signed
2. Female subjects of childbearing potential, defined as not surgically sterile or at least two (2) years postmenopausal, must agree to use one of the following forms of contraception from screening through the last study visit: hormonal (oral, implant, or injection) begun >30 days prior to screening; barrier (condom, diaphragm, or cervical cap with spermicide); intrauterine device (IUD). Acceptable contraceptive options may also include abstinence, relationship with same sex partner or partner who has had a vasectomy at least six (6) months prior to the screening visit
3. Male subjects only: willing to use contraception or abstain from sexual activity beginning with the first exposure to study drug and continuing until discharged from the study due to completion or Early Termination
4. Healthy, as determined by the Investigator, based on medical and dental history, concurrent illnesses, laboratory results, concomitant medications, oral cavity assessment, and targeted physical examination (extraoral, head and neck) during Screening
5. Have a minimum of six unrestored bicuspids and molars with ≤50% of molars and bicuspids having restorations, crowns, sealants or are missing
6. Demonstrated ability to expectorate ≥2mL of stimulated saliva in 5 minutes
7. Have a salivary S. mutans of 1.0 x 10e5 CFUs/mL or greater at Screening using MSB agar plating
8. Willing to refrain from using non-study dentifrice and other non-study oral care products (oral care rinses, fluoride products, etc.) during the study
9. Willing to postpone elective dental procedures (e.g., dental cleanings) between Screening and final post-treatment visit
10. Willing and able to comply with oral hygiene and diet instructions
11. Has dentition adequate for custom dental tray gel application
12. Able to understand and sign the Assent and/or Informed Consent Form prior to initiation of study procedures
13. Able to communicate with the Investigator/study center personnel, understand and comply with the study requirements, and willing to return for protocol-specified visits at the appointed times

Exclusion Criteria:

1. Advanced periodontal disease
2. Active caries lesion(s) within 30 days prior to study drug administration (confirmed by comprehensive caries examination including standard radiographs); Note: Subjects presenting with insipient, non-cavitated lesion(s) are not excluded
3. Medical condition (e.g., artificial heart valve, history of infective endocarditis, cardiac transplant with valvular dysfunction, congenital heart disease or total joint replacement) for which antibiotics are recommended prior to dental visits and/or procedures
4. Pathologic lesions of the oral cavity
5. Full or partial dentures, or orthodontic appliances, e.g., night guards, permanent retainers
6. Use of systemic antibiotics, topical oral antibiotics, or use of other drugs, which in the opinion of the Investigator could influence the study outcome, within 30 days prior to Screening
7. Medical history indicating the woman is pregnant, breastfeeding/ lactating or has a positive urine pregnancy test
8. Participation in a clinical trial or receipt of a non-FDA approved therapy within 30 days prior to study drug administration
9. Prior participation in a C16G2 clinical trial and known to have received C16G2 active gel or mouth rinse
10. Presence of any condition or concurrent illness, which in the opinion of the Investigator, would compromise normal immune function, interfere with the use of study dentifrice and oral care products, or interfere with the ability to comply with study requirements, or jeopardize the safety of the subject or the validity of the study results

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Safety of multiple C16G2 Gel administrations as measured by adverse events | Screening to week 41
  Subjects will be monitored for adverse events throughout the study. At specified clinic visits a targeted physical exam and oral cavity assessment will be performed and vital signs will be taken.

SECONDARY OUTCOMES:
Targeted antimicrobial activity of C16G2 Gel applications as measured by a reduction in Streptococcus mutans in saliva and dental plaque | Microbiology assessments at screeninig, weeks 1, 2, 4, 8, 12, 13, 27, and 41
Total bacteria in saliva and dental plaque post-study drug administration | Total bacteria at weeks 1, 2, 13, 14

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wolff, MD, Principal Investigator — New York University, School of Dentistry
Locations (5):
- United States (5):
  - Indiana University School of Dentistry, Indianapolis, Indiana
  - John F. Pittaway, DMD, Kalispell, Montana
  - New York University College of Dentistry, New York, New York
  - University of Pennsylvania School of Dental Medicine, Philadelphia, Pennsylvania
  - Anthony Henegar, DDS, PA, Irving, Texas